CLINICAL TRIAL: NCT02258113
Title: Measuring of Neuro-visual Functionality With New Human Visual System Device Ocusweep
Brief Title: Measuring of Neuro-visual Functionality With Ocusweep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ocuspecto Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: T109/2014
Record Dates: First submitted 2014-09-30; First posted 2014-10-07 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Visual Impairment
MeSH Terms: conditions — Vision Disorders

ARMS (1):
- LEA numbers, Pelli-Robson, Octopus (Other): Comparable generally used method for measuring visual acuity, contrast sensitivity and visual field.
  Interventions: Device: Ocusweep; Device: Ocusweep OcuRT

INTERVENTIONS:
Device: Ocusweep — A novel reaction-time based visual field device.
Device: Ocusweep OcuRT — Vision based choice reaction time test method

SUMMARY:
The aim of this study is to measure visual acuity, contrast sensitivity and visual field by SAP-method using a novel device Ocusweep compared to currently widely used methods. Addition to that, the aim is to validate a novel perimetry method (Visual Search Test, VST) which is based on reaction times in visual decision- making task, where the subject is allowed to move eyes and where the fixation is verified by the subject himself in contrast to standard automatic perimetry (SAP) where prolonged stationary fixation and external fixation monitoring apparatus is required. Reaction-time based visual field device Ocusweep is compared to generally used SAP methods. Those tests will be done for healthy volunteers and for persons with diagnosed eye or brain disease.

Ocusweep OcuRT vision based choice reaction time test is validated for test repeatability and compared to Trail Making Test (TMT), Useful Field of View (UFOV) and Vienna Test System (VTS) reaction time tests. To evaluate the ability to detect unreliable results, OcuRT test is also done under cognitive load and with instructions to cheat the test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Persons suffering diagnosed eye disease
* Persons suffering diagnosed brain disease

Exclusion Criteria:

* No diabetes
* Only one diagnosed disease

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-11; Primary Completion 2021-12 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | One visit per one patient (1h/visit)
  Visual acuity is measured as logMAR unit at the one visit for each patient using a novel reaction-time based visual field device and comparable method.

SECONDARY OUTCOMES:
Contrast sensitivity | One visit per one patient (1h/visit)
  Contrast sensitivity is measured as logCS unit at the one visit for each patient using a novel reaction-time based visual field device and comparable method.
Reaction time visual field | One visit per one patient (1h/visit)
  Reaction time is measured using a novel reaction-time based visual field device and compared with generally used visual field program.
Vision based choice reaction time | One visit per one test subject (1h/visit)
  Reaction time is measured with Ocusweep OcuRT test three times to asses repeatability of the test. OcuRT reaction time results will be compared to Trail Making Test (TMT), Useful Field of View (UFOV) and Vienna Test System (VTS) reaction time tests. To evaluate the ability to detect unreliable results, OcuRT will also be done under cognitive load and with instructions to cheat the test.

CONTACTS AND LOCATIONS:
Locations (1):
- Ocuspecto Oy, Turku, Finland